CLINICAL TRIAL: NCT04328636
Title: Nebulized Magnesium Sulfate for Treatment of Persistent Pulmonary Hypertension of The Newborn
Brief Title: Nebulized MgSO4 in Persistent Pulmonary Hypertension of Newborn
Acronym: NebMag
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Elsayed Abdelkreem, Lecturer of Pediatrics, Sohag University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NebMag-PPHN Study
Record Dates: First submitted 2020-03-29; First posted 2020-03-31 (Actual); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: Persistent Fetal Circulation; Persistent Pulmonary Hypertension of the Newborn; PPHN
Keywords: neonate; persistent fetal circulation; persistent pulmonary hypertension of the newborn; PPHN; Magnesium Sulfate; Nebulizer; hypoxia
MeSH Terms: conditions — Persistent Fetal Circulation Syndrome; Hypoxia

STUDY DESIGN:
Intervention Model Description: Two groups of neonates with PPHN
  1. NebMag group: receive nebulized magnesium sulfate and intravenous placebo.
  2. IVMag group: receive intravenous magnesium sulfate and nebulized placebo.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Each neonate was assigned a unique identification number. Pharmacy filled the active and placebo preparations in similar containers with sealed code for identification. Participants' families, treating clinicians, nurses, echocardiographers, and data collectors were unaware of group assignment and drug/placebo therapy.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- NebMag (Experimental): Neonates with PPHN receiving nebulized magnesium sulfate and intravenous placebo
  Interventions: Drug: Nebulized Magnesium Sulfate
- IVMag (Active Comparator): Neonates with PPHN receiving intravenous magnesium sulfate and nebulized placebo
  Interventions: Drug: Intravenous Magnesium Sulfate

INTERVENTIONS:
Drug: Nebulized Magnesium Sulfate — Nebulized magnesium sulfate (isotonic solution) 256 mg every 15 minutes
  Arms: NebMag
Drug: Intravenous Magnesium Sulfate — Intravenous magnesium sulfate 200 mg/kg over 30 minutes, followed by a continuous infusion at a rate of 50 mg/kg/hour
  Arms: IVMag

SUMMARY:
The aim of this pilot randomized controlled blinded study is to evaluate the feasibility of using nebulized magnesium sulfate in the treatment of PPHN.

DETAILED DESCRIPTION:
The effectiveness and safety of nebulized magnesium sulfate (using isotonic solution in a dose of 1024 mg/hour) is compared with intravenous magnesium sulfate (200 mg/kg over 30 minutes, followed by 50 mg/kg/hour) in treating mechanically ventilated neonates with severe persistent pulmonary hypertension of the newborn.

ELIGIBILITY:
Inclusion Criteria:

Newborns with PPHN fulfilling the following:

1. born at ≥ 37 weeks gestational age.
2. birth weight between 2.5 and 4 kg.
3. post-natal age between 6 and 72 hours.
4. connected to mechanical ventilation with an oxygenation index (OI) > 30 on two occasions at least 15 minutes apart.
5. documented PPHN confirmed by echocardiography.

Exclusion Criteria:

1. failure to obtain informed consent.
2. infants of mothers who received magnesium sulfate within 48 hours before labor.
3. congenital heart diseases (other than PDA and foramen ovale).
4. major congenital anomalies (including congenital diaphragmatic hernia and lung hypoplasia).
5. prior need for cardiopulmonary resuscitation.
6. mean arterial blood pressure (MABP) < 35 mmHg despite therapy with volume infusions and inotrpic support.
7. impaired kidney function.
8. prior administration of pulmonary vasodilators.

Ages: 6 Hours to 72 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 28 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
Oxygenation index (OI) | At baseline to 2, 6, 12, and 24 hours following study drug administration.
  Change in oxygenation index (OI) calculated by the classic formula:
  OI = [(FiO2 * MAP) / PaO2]
  FiO2 expressed in %; MAP in cmH2O/mmHg; and PaO2 in mmHg

SECONDARY OUTCOMES:
Mean arterial blood pressure (MABP) | At baseline to 2, 6, 12, and 24 hours following study drug administration.
  Changes in mean arterial blood pressure
Serum magnesium level | At baseline to 12 hours after study drug adminstration
  Changes in serum magnesium level
Vasoactive Inotropic Score (VIS) | At baseline to 2, 6, 12, and 24 hours following study drug administration
  Changes in VIS calculated by the classic formula:
  VIS = dopamine dose (µg/kg/min) + dobutamine dose (µg/kg/min) + 100 × epinephrine dose (µg/kg/min) + 100 × norepinephrine dose (µg/kg/min) + 10 × milrinone dose (µg/kg/min) + 10,000 × vasopressin dose (U/kg/min)

CONTACTS AND LOCATIONS:
Overall Officials: Elsayed Abdelkreem, MD, PhD, Principal Investigator — Faculty of Medicine, Sohag University
Locations (1):
- Neonatal Intensive Care Unit, Sohag University Hospital, Sohag, Egypt

REFERENCES:
- [Derived] Abdelkreem E, Mahmoud SM, Aboelez MO, Abd El Aal M. Nebulized Magnesium Sulfate for Treatment of Persistent Pulmonary Hypertension of Newborn: A Pilot Randomized Controlled Trial. Indian J Pediatr. 2021 Aug;88(8):771-777. doi: 10.1007/s12098-020-03643-y. Epub 2021 Jan 8. PMID 33415555